CLINICAL TRIAL: NCT01962961
Title: A Randomized, Placebo-Controlled Pilot Trial Assessing Two Doses of N-Acetylcysteine on Changes in Oxidative Stress and Endothelial Function in HIV-infected Older Adults Receiving Stable Antiretroviral Therapy
Brief Title: N-acetylcysteine to Reduce Oxidative Stress and Improve Endothelial Function in HIV-infected Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: BioAdvantex Pharma (Unknown)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IU SRI 1306011647
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-12

CONDITIONS: HIV; Endothelial Dysfunction; Oxidative Stress
Keywords: HIV; Endothelial function; Oxidative stress; Cardiovascular disease; N-acetylcysteine
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PharmaNAC 1800 mg (Experimental): PharmaNAC 900 mg orally twice daily for 8 weeks
  Interventions: Dietary Supplement: PharmaNAC (N-acetylcysteine); Dietary Supplement: Matching placebo
- PharmaNAC 3600 mg (Experimental): PharmaNAC 1800 mg orally twice daily for 8 weeks
  Interventions: Dietary Supplement: PharmaNAC (N-acetylcysteine)
- Placebo (Placebo Comparator): Matching placebo pills given twice daily for 8 weeks
  Interventions: Dietary Supplement: Matching placebo

INTERVENTIONS:
Dietary Supplement: PharmaNAC (N-acetylcysteine) — PharmaNAC is considered a nutritional supplement and can be obtained without a prescription. All participants will be asked to ingest two tablets twice per day during this trial. For those randomized to PharmaNAC 1800 mg twice daily, this will be two active tablets twice per day. For those randomized to PharmaNAC 900 mg twice daily, this will be one active tablet twice per day and one matching placebo tablet twice per day. For those randomized to placebo, this will be two matching placebo tablets twice per day.
  PharmaNAC can be taken with or without food. The effervescent tablets should be dissolved in 8 oz. of water or juice prior to oral intake. Each participant will take study drug and/or matching placebo for 8 weeks (up to 60 days).
  Other Names: N-acetylcysteine; NAC
  Arms: PharmaNAC 1800 mg; PharmaNAC 3600 mg
Dietary Supplement: Matching placebo — Inactive pill that matches PharmaNAC on taste, color, and appearance.
  Arms: PharmaNAC 1800 mg; Placebo

SUMMARY:
The goal of this study is to determine if n-acetylcysteine, given as PharmaNAC, reduces oxidative stress and improves vascular function in HIV-infected older adults already on HIV treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to compare 8-week changes in circulating levels of malondialdehyde (MDA), circulating levels of F2-isoprostanes, and flow-mediated dilation (FMD) of the brachial artery in older HIV-infected adults already receiving virologically suppressive antiretroviral therapy (ART) who are then randomized to either NAC 900 mg twice daily, NAC 1800 mg twice daily, or placebo. The relative efficacy and safety of these two doses of NAC will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by (1) any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or (2) by two detectable HIV-1 antigens, or (3) two detectable plasma HIV-1 RNA viral loads.
* Age equal to or greater than 50 years.
* Receipt of antiretroviral therapy of any kind for at least 6 months prior to screening.
* HIV-1 RNA level < 75 copies/mL at screening.
* For women who are still of reproductive potential, a negative urine pregnancy test at screening and willingness to use two forms of birth control during the course of the study. Acceptable forms of birth control include condoms (with or without a gel that can kill sperm), a diaphragm or cervical cap (with or without a gel that can kill sperm), an intrauterine device (IUD), or hormonal-based birth control ("the pill").

Exclusion Criteria:

* Inability to complete written, informed consent.
* Incarceration at the time of any study visit.
* Known allergy or intolerance to n-acetylcysteine.
* Use of n-acetylcysteine within 180 days of screening.
* Diagnosed vascular disease (history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease).
* History of congestive heart failure even if currently compensated.
* History of portal hypertension or hepatic cirrhosis (either clinically diagnosed or histologically diagnosed).
* Diagnosed disease or process, besides HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, other collagen vascular diseases).
* Known or suspected malignancy requiring systemic treatment within six months of screening.
* History of ADA-defined diabetes mellitus (115)
* History of migraine headaches.
* History of Raynaud's phenomenon.
* History of cardiac arrhythmias or cardiomyopathy.
* Uncontrolled hyperthyroidism or hypothyroidism, defined as TSH values outside of the local reference range on most recent clinical assessment.
* Asthma or COPD requiring daily use of beta-2-agonist therapy (e.g. albuterol)
* History of carotid bruits.
* Creatinine clearance < 50 mL/min (using the Cockcroft-Gault equation) using a serum creatinine level measured at screening.
* Hemoglobin < 9.0 g/dL at screening.
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) > 3 times ULN at screening.
* Total bilirubin > 2.5 times ULN at screening; if the participant is receiving atazanavir, then s/he would be excluded if total bilirubin is > 3.5 times ULN at screening.
* Therapy for serious medical illnesses within 14 days prior to screening.
* Pregnancy or breastfeeding during the course of the study.
* Uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at screening.
* Receipt of investigational agents, cytotoxic chemotherapy, systemic glucocorticoids (of any dose), or anabolic steroids at screening.
* Previous receipt of stavudine or didanosine for more than 7 cumulative days.
* Receipt of daily Vitamin C or Vitamin E supplements at screening.
* Alcohol intake more than the equivalent of one 8 oz. of wine daily for the 7 days prior to screening.
* Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Health University Hospital, Indiana Clinical Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PharmaNAC 1800 mg: PharmaNAC 900 mg orally twice daily for 8 weeks
  PharmaNAC (N-acetylcysteine): PharmaNAC is considered a nutritional supplement and can be obtained without a prescription. All participants will be asked to ingest two tablets twice per day during this trial. For those randomized to PharmaNAC 1800 mg twice daily, this will be two active tablets twice per day. For those randomized to PharmaNAC 900 mg twice daily, this will be one active tablet twice per day and one matching placebo tablet twice per day. For those randomized to placebo, this will be two matching placebo tablets twice per day.
  PharmaNAC can be taken with or without food. The effervescent tablets should be dissolved in 8 oz. of water or juice prior to oral intake. Each participant will take study drug and/or matching placebo for 8 weeks (up to 60 days).
  Matching placebo: Inactive pill that matches PharmaNAC on taste, color, and appearance.
- PharmaNAC 3600 mg: PharmaNAC 1800 mg orally twice daily for 8 weeks
  PharmaNAC (N-acetylcysteine): PharmaNAC is considered a nutritional supplement and can be obtained without a prescription. All participants will be asked to ingest two tablets twice per day during this trial. For those randomized to PharmaNAC 1800 mg twice daily, this will be two active tablets twice per day. For those randomized to PharmaNAC 900 mg twice daily, this will be one active tablet twice per day and one matching placebo tablet twice per day. For those randomized to placebo, this will be two matching placebo tablets twice per day.
  PharmaNAC can be taken with or without food. The effervescent tablets should be dissolved in 8 oz. of water or juice prior to oral intake. Each participant will take study drug and/or matching placebo for 8 weeks (up to 60 days).
Period: Overall Study
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo
Started | 9 | 8 | 7
Completed | 9 | 7 | 6
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 7 | 24
Age, Continuous [Mean (Full Range); unit: years] | 52 [50 to 61] | 53 [51 to 57] | 54 [50 to 57] | 53 [50 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 8 | 8 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 8 | 8 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 4 | 13
  White | 1 | 5 | 3 | 9
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Circulating Malondialdehyde Levels
Description: Measure of oxidative stress
Time Frame: Baseline and 8 weeks
Population: Analysis population includes those who completed the 8 week trial and had both baseline and week 8 values available.
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo
Number analyzed (Participants) | 9 | 7 | 6
micromolar | 0.17 (1.74) | -0.12 (.054) | -0.00 (0.56)

2. Primary Outcome: Change in Circulating F2-isoprostane Levels
Description: Oxidative stress measure
Time Frame: Baseline and 8 weeks
Population: Analysis population includes those who completed the 8 week trial and had both baseline and week 8 values available.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo
Number analyzed (Participants) | 9 | 7 | 6
pg/mL | -12.78 (26.39) | -4.84 (28.85) | 11.76 (28.76)

3. Primary Outcome: Change in Flow-mediated Dilation (FMD) of the Brachial Artery
Description: Measure of endothelial function
Time Frame: Baseline and 8 weeks
Population: Analysis population includes those who completed the 8 week trial and had both baseline and week 8 values available.
Measure: Mean (Standard Deviation); unit: Percentage of vessel diameter
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo
Number analyzed (Participants) | 7 | 9 | 6
Percentage of vessel diameter | 0.51 (2.00) | -.046 (2.18) | -1.15 (2.56)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | PharmaNAC 1800 mg | PharmaNAC 3600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 6/9 | 6/8 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PharmaNAC 1800 mg (N=9) | PharmaNAC 3600 mg (N=8) | Placebo (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Increased HIV viral load (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Urinary infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion/sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No